CLINICAL TRIAL: NCT06486428
Title: A Study to Evaluate a Remote, Decentralized, Direct-to-Patient Strategy for Clinical Research Engagement of Patients With Small Cell Lung Cancer (SCLC).
Brief Title: Small Cell Lung Cancer Community Engagement to Eliminate Research Discepancies
Acronym: SUCCEED
Status: Recruiting | Type: Observational
Sponsor: Addario Lung Cancer Medical Institute (Other)
Responsible Party: Sponsor
Other Study IDs: ALCMI-023
Record Dates: First submitted 2023-12-15; First posted 2024-07-03 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Small-cell Lung Cancer
Keywords: SCLC; Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Two (2) EDTA tubes of whole blood (approx 10 mL per tube) will be sent to the ALCMI biobank for processing and storage (baseline and at month 3).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SCLC (primary de novo): Blood collection, survey (baseline and Month 3)
- SCLC (transformed): Blood collection, survey (baseline and Month 3)

SUMMARY:
This study will evaluate if a direct-to-patient, de-centralized, remote approach will improve clinical research outreach and engagement for patients with SCLC, in the context of a bio-specimen collection study. The study will also assess self-reported preferences and needs of patients with SCLC, regarding choosing and accessing novel therapies in research or standard clinical care settings and supportive gaps in this area, through an initial and 3 month follow up survey.

DETAILED DESCRIPTION:
This is a non-interventional, non-treatment, non-randomized, single coordinating center, study to determine the feasibility of decentralized bio-specimen collection in USA-based adult subjects with SCLC, to be conducted in conformance with Good Clinical Practices. Potential study subjects will be referred to contact staff through a dedicated study webpage form or dedicated study phone hotline at the coordinating center (ALCMI) who will handle informed consent, coordinate remote blood sample collection with study subjects, and collect medical records to confirm diagnosis and treatment history. Subjects will also be asked to complete a baseline and follow up questionnaire/survey documenting their self-report diagnosis, treatment history, factors impacting care and quality of life, and needs/preferences regarding supportive resources.

Patients who have been diagnosed with either extensive stage primary SCLC or patients diagnosed with primary NSCLC who experienced histological "transformation" with a SCLC component after initial diagnosis and subsequent treatment (transformed SCLC; tSCLC) will be invited to volunteer for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women greater than or equal to 18 years of age at the time of consent
2. Ability to read, write and communicate in English
3. Provide voluntary consent to participate in this study, documented via a signed informed Consent Form (ICF)
4. Willing to provide clinical and medical information related to his/her cancer diagnoses to the study team as required
5. Willing to comply with the requirements of the study
6. Diagnosis of extensive stage primary SCLC or tSCLC

Exclusion Criteria:

1. Known existence of an uncontrolled intercurrent illness including, but not limited to, psychiatric illness or social situations that would impair compliance with study requirements
2. Subjects who previously enrolled to this study

Note: Concurrent enrollment in other clinical trials is NOT exclusionary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (USA-based) with a diagnosis of extensive stage primary SCLC or tSCLC
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of conducting trial in SCLC population | 12 months
  Percentage of overall eligible subjects enrolled. Percentage of primary SCLC eligible subjects enrolled. Percentage of tSCLC eligible subjects enrolled. Percentage of SCLC eligible subjects enrolled compared to percentage of tSCLC eligible subjects enrolled. Percentage of primary SCLC enrolled subjects completed. Percentage of tSCLC enrolled subjects completed. Percentage of SCLC enrolled subjects completed compared to percentage of tSCLC enrolled subjects completed. Overall reasons for early termination. Reasons for early termination from trial in primary SCLC enrolled. Reasons for early termination from trial in tSCLC enrolled.

OTHER OUTCOMES:
Bio-specimen collection | 12 months
  Percentage of blood collections during trial in overall enrolled and in SCLC enrolled compared to in tSCLC enrolled.
  Reasons for failure to obtain blood collections. Percentage of successful blood collections during trial (Overall and in SCLC compared to tSCLC).
  Reasons for failure to obtain blood collections. Percentage of successful blood collections during trial (Overall and in SCLC compared to tSCLC). Reasons for failure to obtain blood collections.
Subject Surveys (baseline and at 3 months) | 3 months
  Percentage of successful Survey completions; at baseline; at Month 3. Reasons for failure to complete Survey(s).

CONTACTS AND LOCATIONS:
Overall Officials: Christine Lovly, MD PhD, Principal Investigator — Vanderbilt-Ingram Cancer Center, Nashville, TN
Locations (52):
- United States (52):
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Alabama
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Alaska
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Arizona
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Arkansas
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, California
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Colorado
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Connecticut
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Delaware
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, District of Columbia
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Florida
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Georgia
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Hawaii
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Idaho
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Illinois
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Indiana
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Iowa
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Kansas
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Kentucky
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Louisiana
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Maine
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Maryland
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Massachusetts
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Michigan
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Minnesota
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Mississippi
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Missouri
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Montana
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Nebraska
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Nevada
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, New Hampshire
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, New Jersey
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, New Mexico
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, New York
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, North Carolina
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, North Dakota
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Ohio
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Oklahoma
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Oregon
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Pennsylvania
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Rhode Island
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, South Carolina
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, South Dakota
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Texas
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Utah
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Vermont
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Virginia
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Washington
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, West Virginia
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Wisconsin
  - Https://Alcmi.Org/Clinical-Trials/Current-Studies/Succeed-Study.Html, Multiple Locations, Wyoming

IPD SHARING:
Plan to Share IPD: No